CLINICAL TRIAL: NCT05602870
Title: Acceptability of Advanced Chronic Liver Disease Screening by Transient Elstography (Fibroscan ®) in Patients Hospitalised in Psychiatric Unit: a Single Center Prospective Study
Brief Title: Advanced Chronic Liver Disease Screening by Transient Elstography in Patients Hospitalised in a Psychiatric Unit
Acronym: HEPSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL22_0114
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Psychiatric Disorder; Psychiatric Hospitalization; Advanced Chronic Liver Disease; Liver Fibrosis
Keywords: psychiatric disorders; advanced liver disease; alcoholic liver diseases; viral hepatitis; transient elastography (Fibroscan ®)
MeSH Terms: conditions — Mental Disorders; Liver Cirrhosis; Liver Diseases, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychiatric patient (Experimental): All patients having psychiatric disorders and hospitalised in a Psychiatry Unit of CHU Montpellier will have an non invasive evaluation of liver fibrosis after giving their consent
  Interventions: Diagnostic Test: non invasive evaluation of liver fibrosis by transient elastography (Fibroscan ®)

INTERVENTIONS:
Diagnostic Test: non invasive evaluation of liver fibrosis by transient elastography (Fibroscan ®) — A Fibroscan will be performed and the result will be given to the patient. A follow-up will be organized in the event of a diagnosis of severe fibrosis. If the serologies for hepatitis B and C cannont be recovered, patient will be able to benfit from a rapid diagnostic orientation test (TROD) (minimally invasive capillary venous sampling at the fingertip) for these 2 serologies.

SUMMARY:
Scares data exists concerning the prevalence of chronic liver diseases in people with psychiatric disorders.

There are still many barriers to screening and linkage to care for patients having somatic illness.

Moreover follow-up of these patients may be difficult because of poor access to care, sometimes marginalization, and insufficient compliance with health programs.

The aim of this study is to asses acceptability of of advanced chronic liver disease screening by transient elstography (Fibroscan ®) in patients hospitalised in a psychiatric unit.

DETAILED DESCRIPTION:
Scares data exists concerning the prevalence of chronic liver diseases in people with psychiatric disorders.

There are still many barriers to screening and linkage to care for patients having somatic illness.

Moreover follow-up of these patients may be difficult because of poor access to care, sometimes marginalization, and insufficient compliance with health programs.

Transient elastography is a useful tool validated for early diagnosis advanced chronic liver disease.It is non-invasive, fast, and gives immediate results.

The aim of this study is to assess acceptability of of advanced chronic liver disease screening by transient elstography (Fibroscan ®) in patients hospitalised in psychiatric unit.

Moreover, we will estimate de prevalence of advanced chronic liver diseases according to specific causes in psychiatry unit We hypothesize that the fact of offering psichiatric patents a non-invasive analysis of hepatic fibrosis will improve the detection of serious liver diseases and linkage to care.

ELIGIBILITY:
Inclusion criteria

* adults ≥18 years
* having a psychiatric condition and hospitalized in a psychiatry unit of CHU Montpellier , France
* patients who lack capacity of consent if legal representative consents
* involuntary psychiatric hospitalization, if consent is given

Exclusion criteria

* lack of written consent
* Unable to understand nature and objective of the methodology
* Pregnant or breast feeding woman
* Not affiliated with a French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
acceptability of non invasive assessement of liver fibrosis by Fibroscan in psychiatric patients | At Inclusion
  Number of patient who have agreed to do fibroscan screening among patient to whom it was offered.

SECONDARY OUTCOMES:
Prevalence of advanced liver disease in psychiatric patients | At inclusion
  Number of patient who are diagnosed with advanced liver disease among patient to whom it was offered.
prevalence of excessive alcohol or drug consumption in psychiatric patients | At inclusion
  Number of patient with excessive alcohol/drug consumption
prevalence of passed or active drug consumption (intraveinous, inhaled or sniffed) in psychiatric patients | At Inclusion
  Number of patient with excessive alcohol/drug consumption
prevalence of viral hepatitis in psychiatric patients | At Inclusion
  Number of patient diagnosed with viral hepatitis B, D, C
correlation between advanced chronic liver diseases and risk factors for liver diseases in psychiatric patients | 1 to 3 month after inclusion
  Number of patients with advanced chronic liver disease among those having risk factors for chronic liver disease
assessment of referral to medical care when advanced fibrosis was diagnosed, regardless of its etiology | 1 to 3 month after inclusion
  Number of patients that have actually came to their medical appoint after advanced fibrosis diagnosis
reason for refusal of non invasive evaluation of chronic liver disease | At Inclusion
  rate of reasons of refusal according to reason of hospitalization, sector, duration of hospitalization, time spend in study explaination, patient reflection time

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France